CLINICAL TRIAL: NCT00273169
Title: Use of the PSA 4000 Monitor in the Post-Operative Period in Patients Undergoing Major Surgery
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Other Study IDs: 110-05
Record Dates: First submitted 2006-01-06; First posted 2006-01-09 (Estimated); Last update posted 2010-01-15 (Estimated); Status verified 2010-01

CONDITIONS: Postoperative

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Evaluate correlation between the values from the PSA monitor and clinical assessment of sedation with the RASS on postoperative patients.

DETAILED DESCRIPTION:
Assessing level of sedation in critically ill patients is an integral part of intensive care practice. Sedation scales, such as the Richmond Agitation-Sedation Score (RASS) 1, have been developed, but are imperfect in a general population and of limited use when muscle relaxants are administered. Instruments have been developed to examine cerebral electrical activity using processed EEG in an attempt to determine state of awareness.2 The Bispectral Index (BIS) is a statistically derived measure of cerebral electrical activity to assess cortical-subcortical interaction. The BIS was determined by repeated studies on patients anesthetized in the operating room (OR) with the assumption that sedation is associated with a lack of awareness and recall.2 The Patient State Analyzer (PSA 4000) is a 4-channel processed EEG reading using an advanced algorithm that interprets changes in regional brain activity providing a numerical assessment (ranging from 0-100; 0 = no central nervous system [CNS] activity, 100 = awake) to assess the degree of sedation. The PSA 4000 (PSA) is an advancement over the BIS monitor as the BIS is a single channel whereas the PSA is a 4-channel monitor. Additionally, the PSA monitor has new proprietary software for analysis of the EEG data. The PSA is relatively new and thus there is little published data to evaluate its use in the operating room (OR) or the intensive care unit (ICU).

ELIGIBILITY:
Detailed Population Description: The study population will include those patients that have undergone surgery under general anesthesia at St. Marys Hospital, Mayo Clinic Rochester, admitted to the 7MB D/E Intensive Care Unit and require intubation and mechanical ventilation for a period of at least 4 hours after admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Detailed Population Description: The study population will include those patients that have undergone surgery under general anesthesia at St. Marys Hospital, Mayo Clinic Rochester, admitted to the 7MB D/E Intensive Care Unit and require intubation and mechanical ventilation for a period of at least 4 hours after admission
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2005-07; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francis X. Whalen, Jr., M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States